CLINICAL TRIAL: NCT01777347
Title: 3% Hypertonic Saline to Reduce Hospitalization Rate in Acute Viral Bronchiolitis: a Randomized Double Blind Clinical Trial
Brief Title: Efficacy of 3% Hypertonic Saline in Acute Viral Bronchiolitis
Acronym: GUERANDE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IDRCB 2012-A00228-35; P110143 (Other: AP-HP); AOM11036 (Other: AP-HP)
Record Dates: First submitted 2012-11-14; First posted 2013-01-28 (Estimated); Last update posted 2014-07-28 (Estimated); Status verified 2014-07

CONDITIONS: Acute Viral Bronchiolitis
Keywords: Keywords provided by ASSISTANCE PUBLIQUE HOPITAUX DE PARIS:; Acute Viral bronchiolitis; Hypertonic saline; Hospitalization; Infants; Hospital admissions; Additional relevant MeSH terms:; Bronchiolitis; Bronchiolitis, Viral; Bronchial Diseases; Respiratory Tract Diseases; Lung Diseases, Obstructive; Respiratory Tract Infections; Virus Diseases
MeSH Terms: conditions — Bronchiolitis; Bronchiolitis, Viral; Bronchial Diseases; Respiratory Tract Diseases; Lung Diseases, Obstructive; Respiratory Tract Infections; Virus Diseases | interventions — Sodium Chloride; Saline Solution, Hypertonic; Inhalation; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 3% Saline (Experimental): Nebulized 3% Saline
  Interventions: Drug: 3% Saline
- 0.9% Normal Saline (Placebo Comparator): Nebulized 0.9% normal saline
  Interventions: Drug: 0.9% Normal Saline

INTERVENTIONS:
Drug: 3% Saline — Two 4 mL nebulization of 3% saline with 20 minutes interval
  Other Names: 3% Hypertonic Saline Solution for Inhalation (Mucoclear 3%)
  Arms: 3% Saline
Drug: 0.9% Normal Saline — Two 4 mL nebulization of 0.9% normal saline with 20 minutes interval
  Other Names: 0.9% Saline Solution for Inhalation
  Arms: 0.9% Normal Saline

SUMMARY:
The purpose of this study is to determine whether nebulized hypertonic saline solution reduces the admission rate 48 hours after initial treatment in the emergency department, when compared to normal saline solution (control).

DETAILED DESCRIPTION:
Acute viral bronchiolitis remains a significant cause of hospitalization and to date, no treatment reduce the rate of hospitalization. The only accepted treatment for bronchiolitis is nasal cleaning, hydration and for hospitalized hypoxemic infants, oxygen administration.

Several studies shown that nebulization of hypertonic saline solution reduce length of stay in hospital for hospitalized infant but effect on rate of hospitalization remains unclear.

The investigators propose a randomized double blind multicenter clinical trial on infants 6 weeks to 12 months old with moderate or severe bronchiolitis, in 21 emergency departments of hospitals situated France, during 2 winter seasons.

The investigators hypothesize that infants with bronchiolitis treated with nebulized hypertonic 3% saline solution would have less risk of being hospitalized. Our principal objective is to determine if nebulized 3% hypertonic saline solution reduces admission rate 24 hours after treatment compared to placebo.

Secondary objectives are to compare between groups intensity of respiratory symptoms measured by RDAI clinical score, duration of symptoms, length of hospital stay for hospitalized infants, adverse effects and health care utilization.

Patients presenting to the Emergency Department with a diagnosis of moderately severe bronchiolitis will be approached for entry into the study. After the initial routine assessment, informed consent will be obtained and the infant will be randomized to receive treatment in a double-blinded fashion 4 ml of nebulized study solution either 3% hypertonic saline (HS, study group) or 0.9% saline (NS, control group) every 20 minutes for a total of 2 doses. After an observation period of 20 minutes following the last dose, the infant will be reassessed by the attending physician in the ER for disposition (admit, discharge home). All subsequent therapy, if needed, will be at the sole discretion of the attending physician. The family of each recruited subject will be contacted by phone 2, 7, 14 and 28 days later to assess resolution of symptoms.

Clinical response to the above treatment will also be determined independently by the study physician utilizing a standardized respiratory scoring system, the Respiratory Distress Assessment Instrument (RDAI), at study entry and after each nebulization. The primary outcome measure is the rate of admission to hospital between the study and control groups 24 hours after inclusion. Secondary outcomes measure will involve the assessment of change in the RDAI between study entry and post-treatment, adverse effects, length of stay for hospitalized infant and health care utilization.

ELIGIBILITY:
Inclusion Criteria:

* Age 6 weeks through 12 months
* First moderate to severe episode of acute viral bronchiolitis (history of viral upper respiratory tract infection plus wheezing and/or crackles on chest auscultation with respiratory distress ).
* Admission in Emergency Department
* Parental/guardian permission (informed consent)

Exclusion Criteria:

* prematurity < 37 weeks
* artificial ventilation in the neonatal period
* Chronic lung or heart disease
* history of immunodeficiency
* past use of nebulized HS
* initial need for intensive care of assisted ventilation
* Non-French speaking parent/guardian

Ages: 6 Weeks to 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 778 (Actual)
Dates: Start 2012-10; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Admission rate | 24 hours

SECONDARY OUTCOMES:
change in RDAI score | 2 hours
Number of Participants with Adverse Events | 2 hours
length of hospitalization for hospitalized infant | 1 month
health care utilisation | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Vincent Gajdos, MD, PhD, Principal Investigator — Assistance Publique Hôpitaux de Paris - Paris Sud Medical School
Locations (21):
- France (21):
  - Hôpital Jean Verdier, Bondy
  - Hôpital Ambroise Paré, Boulogne
  - CHU, Caen
  - Hôpital Antoine Béclère, Clamart
  - Hôpital Louis Mouriez, Colombes
  - Centre Hospitalier Sud Francilien, Corbeil
  - Centre Hospitalier intercommunal de Créteil, Créteil
  - Centre Hospitalier de Fontainebleau, Fontainebleau
  - Hôpital Kremlin Bicêtre, Le Kremlin-Bicêtre
  - Hôpital Jeanne de Flandre, Lille
  - Hôpital Hôpital Mère Enfants, Limoges
  - Hôpital Hôpital Femme Mère Enfants, Lyon
  - Hôpital Nord, Marseille
  - Hôpital d'enfants, Nancy
  - Hôpital Mère - Enfants, Nantes
  - CHU Lenval, Nice
  - Hôpital Necker-Enfants Malades, Paris
  - Hôpital Robert Debré, Paris
  - Hôp Charles Nicolle - CHU Rouen, Rouen
  - Hôpital des enfants, Toulouse
  - André Mignot, Versailles

REFERENCES:
- [Derived] Angoulvant F, Bellettre X, Milcent K, Teglas JP, Claudet I, Le Guen CG, de Pontual L, Minodier P, Dubos F, Brouard J, Soussan-Banini V, Degas-Bussiere V, Gatin A, Schweitzer C, Epaud R, Ryckewaert A, Cros P, Marot Y, Flahaut P, Saunier P, Babe P, Patteau G, Delebarre M, Titomanlio L, Vrignaud B, Trieu TV, Tahir A, Regnard D, Micheau P, Charara O, Henry S, Ploin D, Panjo H, Vabret A, Bouyer J, Gajdos V; Efficacy of 3% Hypertonic Saline in Acute Viral Bronchiolitis (GUERANDE) Study Group. Effect of Nebulized Hypertonic Saline Treatment in Emergency Departments on the Hospitalization Rate for Acute Bronchiolitis: A Randomized Clinical Trial. JAMA Pediatr. 2017 Aug 7;171(8):e171333. doi: 10.1001/jamapediatrics.2017.1333. Epub 2017 Aug 7. PMID 28586918